CLINICAL TRIAL: NCT01590225
Title: A Phase 3 Study to Assess the Efficacy and Safety of Boceprevir in Combination With Peginterferon Alfa-2b Plus Ribavirin in Pediatric Subjects With Chronic Hepatitis C Genotype 1
Brief Title: Efficacy and Safety of Boceprevir in Combination With Peginterferon Alfa-2b Plus Ribavirin in Pediatric Subjects With Chronic Hepatitis C Genotype 1 (P08034)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P08034; 2010-024260-17 (EudraCT Number)
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A: boceprevir + peginterferon alpha-2b + ribavirin (Experimental)
  Interventions: Drug: Boceprevir; Drug: Peginterferon alpha-2b; Drug: Ribavirin
- Part B: boceprevir + peginterferon alpha-2b + ribavirin (Experimental)
  Interventions: Drug: Boceprevir; Drug: Peginterferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Drug: Boceprevir — Boceprevir will be administered orally at a dose of 11.4 mg/kg three-times daily (TID) for 24 weeks. The boceprevir dose will be calculated based on 11.4 mg/kg and will then be rounded to the nearest 200-mg value for subjects in the oldest age group, or to the nearest 100-mg or 200-mg value for the subjects in the two youngest age groups.
  Other Names: Victrelis®; SCH 503034
  Arms: Part A: boceprevir + peginterferon alpha-2b + ribavirin
Drug: Peginterferon alpha-2b — Peginterferon alpha-2b will be administered subcutaneously at a dose of 60 μg/m^2 once weekly (QW) for 24 weeks.
  Other Names: Pegintron®; Sylatron®
  Arms: Part A: boceprevir + peginterferon alpha-2b + ribavirin
Drug: Ribavirin — The dose of ribavirin will be approximately 15 mg/kg/day administered orally in two divided doses (twice daily [BID]) for 24 weeks.
  Other Names: Copegus®; Rebetol®; RibaTab®; Ribasphere®
  Arms: Part A: boceprevir + peginterferon alpha-2b + ribavirin
Drug: Boceprevir — Boceprevir will be administered orally at a dose of 11.4 mg/kg three-times daily (TID) for up to 48 weeks. The boceprevir dose will be calculated based on 11.4 mg/kg and will then be rounded to the nearest 200-mg value for subjects in the oldest age group, or to the nearest 100-mg or 200-mg value for the subjects in the two youngest age groups.
  Arms: Part B: boceprevir + peginterferon alpha-2b + ribavirin
Drug: Peginterferon alfa-2b — Peginterferon alpha-2b will be administered subcutaneously at a dose of 60 μg/m^2 once weekly (QW) for 48 weeks.
  Other Names: Pegintron®; Sylatron®
  Arms: Part B: boceprevir + peginterferon alpha-2b + ribavirin
Drug: Ribavirin — Drug: Ribavirin
  The dose of ribavirin will be approximately 15 mg/kg/day administered orally in two divided doses (twice daily [BID]) for 48 weeks.
  Other Names: Copegus®; Rebetol®; RibaTab®; Ribasphere®
  Arms: Part B: boceprevir + peginterferon alpha-2b + ribavirin

SUMMARY:
This is a three-part (Part A, Part B, and Part C), open-label, multicenter study of boceprevir in pediatric participants with chronic hepatitis C (CHC) genotype 1 (GT1). In Part A and Part B, efficacy and safety will be evaluated in participants with CHC GT1 who are non-cirrhotic, treatment naïves (Part A) or who are non-cirrhotic, treatment failures to (peg)interferon/ribavirin or who are cirrhotics (whether treatment naïve or treatment failure) (Part B). Part C is long-term follow up and no study treatment will be administered during this period, but participants who do not achieve viral clearance will be allowed to receive other treatments for CHC.

ELIGIBILITY:
Inclusion Criteria:

* CHC GT1 infection for at least 6 months with with HCV-RNA ≥10,000 IU/mL.
* Treatment naive, non-cirrhotic participants will be eligible for inclusion in Study Part A
* Non-cirrhotic subjects who failed previous (peg)interferon/ribavirin treatment for CHC and cirrhotics, whether treatment naive or treatment failure, will be eligible for inclusion in Study Part B
* To participate in Study Part C, participants must have completed the required post-treatment follow-up in Study Part A or Part B
* Weight ≥ 10 kg to ≤ 125 kg
* Body surface area (BSA) ≥0.46 m^2 and ≤2.5 m^2
* Previous liver biopsy with histology consistent with chronic hepatitis C and no other etiology within 2 years of the screening visit
* Participants with bridging fibrosis or cirrhosis must have an ultrasound within 6 months of the screening visit or between the screening visit and Day 1 with no findings suspicious for hepatocellular carcinoma
* Participant must be able to adhere to dose and visit schedules

Exclusion Criteria:

* Known co-infection with the the human immunodeficiency virus (HIV) or hepatitis B virus (HBsAg positive)
* For Study Part A, participant received any prior hepatitis C treatment, including herbal remedies, with known hepatotoxicity
* For Study Part B, participant received treatment with ribavirin within 90 days or any interferon alpha within 30 days prior to screening
* For Study Part B, participant received previous treatment with a hepatitis C virus protease inhibitor (excepting participants in study P07614, Pharmacokinetics of Boceprevir in Pediatric Subjects With Chronic Hepatitis C Genotype 1)
* For Study Part B, participant required discontinuation of previous (peg)interferon/ribavirin therapy for an adverse event considered by the investigator to be related to (peg)interferon and/or ribavirin
* For Study Part B, participant is currently taking any antiviral/immunomodulatory treatment for hepatitis C
* Participant has taken any investigational drugs, except boceprevir
* Participant has received any of the following medication(s) within 2 weeks prior to the Day 1 visit: midazolam, pimozide, amiodarone, flecainide,

propafenone, quinidine, and ergot derivatives (dihydroergotamine, ergonovine,

ergotamine, methylergonovine)

* Participation in any other clinical trial within 30 days of enrollment or

intent to participate in another clinical trial during participation in the current study

* Evidence of decompensated liver disease
* Child Pugh score >6 (class B and C)
* History of diabetes or hypertension or was born prior to 32 weeks

of gestation and has clinically significant ocular examination findings

* Pre-existing clinically significant psychiatric condition(s)
* Clinical diagnosis of substance abuse
* Any pre-existing medical condition that could interfere with participation in and completion of the study
* Evidence of active or suspected malignancy
* Females who are pregnant, nursing, or intend to become pregnant during

the study period

* Allergy or sensitivity to the investigational products or excipients

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-01-28 (Actual); Primary Completion 2021-08-18 (Estimated); Study Completion 2021-08-18 (Estimated)

PRIMARY OUTCOMES:
Participants Achieving Sustained Viral Response (SVR) at Follow-Up Week 24 in Study Part A | Follow-Up Week 24
Participants Achieving SVR at Follow-Up Week 24 in Study Part B | Follow-Up Week 24
Time to Viral Relapse in Study Part C | Follow-Up Week 24 to 5 Years

SECONDARY OUTCOMES:
Proportion of Participants With Alanine Aminotransferase (ALT) Normalization in Study Part A | Week 2, Week 4, Week 8, Week 12
Participants With Early Virologic Response in Study Part A | Week 2, Week 4, Week 8, Week 12
Proportion of Participants With Undetectable Hepatitis C Virus Ribonucleic Acid (HCV-RNA) in Study Part A | Week 12, End of Treatment, Follow-Up Week 24
Proportion of Participants With Undetectable HCV-RNA Who Also Achieved SVR in Study Part A | Follow-Up Week 12
Proportion of Participants With Alanine Aminotransferase (ALT) Normalization in Study Part B | Week 2, Week 4, Week 8, Week 12
Proportion of Participants With Undetectable HCV-RNA in Study Part B | Week 24, End of Treatment, Follow-Up Week 12
Proportion of Participants With Undetectable HCV-RNA Who Also Achieved SVR in Study Part B | Follow-Up Week 12
Number of Participants Experiencing Treatment-Emergent Adverse Events (AEs) in Study Part A | Week 1 to Follow-Up Visit 24
Number of Participants Experiencing Treatment-Emergent Treatment-Related AEs in Study Part A | Week 1 to Follow-Up Week 24
Number of Participants Experiencing Serious AEs (SAEs) in Study Part A | Week 1 to Follow-Up Week 24
Participants Discontinuing Treatment Due to AEs in Study Part A | Week 1 to Follow-Up Week 24
Change from Baseline in Participant Laboratory Values in Study Part A | Baseline to Follow-Up Week 24
Change From Baseline in Participant Vital Signs in Study Part A | Baseline to Follow-Up Week 24
Number of Participants Experiencing AEs in Study Part B | Week 1 to Follow-Up Week 24
Number of Participants Experiencing SAEs in Study Part B | Week 1 to Follow-Up Week 24
Change from Baseline in Participant Laboratory Values in Study Part B | Week 1 to Follow-Up Week 24
Change From Baseline in Participant Vital Signs in Study Part B | Week 1 to Follow-Up Week 24
Number of Participants Discontinuing From Study Treatment Due to AEs in Study Part B | Week 1 to Follow-Up Week 24